CLINICAL TRIAL: NCT06747234
Title: Effect of Oat Bran Supplementation on Plasma Lipid, Selected Fecal Bacteria, and Short-chain Fatty Acids Receptors Gene Expression in Peripheral Blood Mononuclear Cells in Patients With Coronary Artery Disease
Brief Title: Oat Bran and Plasma Lipid and Fecal Bacteria in Coronary Artery Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 43012538
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Coronary Arterial Disease (CAD)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oat bran (Experimental): Daily consumption of oat bran along with standard medical treatment
  Interventions: Other: Oat bran group
- Control (Other): Standard medical treatment
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Oat bran group — Patients consume 28 grams of oat bran daily for two months in addition to their usual medical treatment.
  Arms: Oat bran
Other: Control (Standard treatment) — Patients receive standard medical treatment.
  Arms: Control

SUMMARY:
The development of atherosclerosis is significantly influenced by the interplay between lipid and inflammatory factors. Endotoxemia, defined as the presence of endotoxins, particularly lipopolysaccharides (LPS) derived from Gram-negative bacteria, in the bloodstream, is closely associated with low-grade inflammation. This chronic, systemic inflammatory response does not reach the severity of acute inflammation but can contribute to the development of atherosclerosis and cardiovascular disease (CVD). Lipopolysaccharide-binding protein (LBP) is a soluble acute-phase protein that binds to bacterial LPS. Elevated levels of LBP have been linked to increased low-grade inflammation, which further exacerbates chronic inflammation and metabolic dysregulation. Dietary fiber, such as oat bran, may have a role in mitigating the effects of endotoxemia and its associated inflammation. Furthermore, dietary fiber could play a role in improving plasma lipid profiles. The present study will investigate the effect of oat bran supplementation on cardiometabolic risk markers, LBP concentrations, selected fecal bacteria, and short-chain fatty acids receptors gene expression in peripheral blood mononuclear cells in patients with coronary artery disease.

DETAILED DESCRIPTION:
As stated by the World Health Organization, cardiovascular diseases (CVDs), particularly coronary artery disease (CAD), represent the primary cause of mortality globally. Atherosclerosis, the primary pathophysiological mechanism underlying CAD, is a multifactorial process, with lipids and inflammatory factors playing a pivotal role. One potential cause of chronic inflammation is endotoxemia, which is a condition resulting from the absorption of lipopolysaccharide (LPS) into the circulatory system. LPS is an active component of the cell wall of gram-negative bacteria derived from the gut microbiota and a potent activator of the innate immune system via the toll-like receptor 4 pathway. The entry of LPS into the systemic circulation ultimately results in the intracellular transcription of several inflammatory mediators, which subsequently trigger an inflammatory response. This is recognized as a contributing factor in the development and progression of atherosclerosis and subsequent coronary artery disease. The presence of bacterial 16S ribosomal RNA belonging to the Enterobacterial family has been identified in atherosclerotic plaques. The protein that binds to LPS in the blood is known as LBP (lipopolysaccharide-binding protein). Serum levels of LBP have been demonstrated to be elevated in patients with angiographically confirmed CAD in comparison to individuals without coronary atherosclerosis.

An increase in dietary fiber intake has the potential to influence plasma lipid components, including LDL cholesterol, HDL cholesterol, and triglycerides. Furthermore, dietary fiber has the potential to influence the composition of the gut microbiota, which may, in turn, influence the levels of LBP and other microbially produced factors, and consequently, cardiovascular health. It has been demonstrated that dietary fiber can facilitate the growth of a more diverse gut microbiota, which in turn produces metabolites that are capable of modulating local and systemic inflammation. Moreover, the impact of a diet rich in fiber on the structure and function of the gut microbiota and the metabolites produced by this microbial community may prove effective in preventing certain CVDs by reducing local and systemic inflammation.

Dietary fiber is metabolized by intestinal bacteria, resulting in the production of metabolites that are subsequently absorbed by intestinal cells. Short-chain fatty acids (SCFAs), including acetate, propionate, and butyrate, are produced by the intestinal microbiota in the large intestine through fermentation of dietary fiber. Research has demonstrated that they function as ligands for a particular group of G protein-coupled receptors, including GPR43 and GPR109A, which are expressed on a range of cells, including white blood cells. The binding of SCFAs to these receptors results in the induction of intracellular signaling, which in turn triggers a wide range of cellular and tissue effects that may be involved in the regulation of metabolism and inflammation. These effects may contribute to the cardioprotective effects of SCFAs.

The present study will investigate the effect of oat bran supplementation on plasma lipid, insulin, inflammatory markers, LBP concentrations, selected fecal bacteria, and short-chain fatty acids receptors gene expression in peripheral blood mononuclear cells in patients with coronary artery disease.

This study employs a randomized controlled clinical trial design without blinding. In this study, patients meeting the eligibility criteria and referred to the Shahid Modarres Medical and Research Center will be selected. The objectives and methodology of the study will be fully explained to them, and written consent will be obtained from all volunteers. The medical records of the patients will be utilized to collate data pertaining to the disease, the pharmacological agents employed, and other pertinent medical information. The study will include measurements of weight and calculation of body mass index (BMI) for all patients at the outset and conclusion of the study. The level of physical activity will be gauged using a physical activity questionnaire at the outset and conclusion of the study. Patients will be randomly assigned to one of two study groups, namely the control group and the oat bran group. The study will be conducted over a period of two months. The control group will receive general dietary advice, including recommendations to reduce saturated fat, sodium, and simple sugar intake. In the oat bran group, in addition to the aforementioned recommendations, patients will consume 28 grams of oat bran per day. All patients will be instructed to refrain from using over-the-counter herbal medicines, probiotic food products (such as yogurt), and probiotic supplements throughout the course of the study.

To assess biochemical blood parameters at the outset and conclusion of the study, a 6 cc venous blood sample will be obtained from all patients via the brachial vein after 12-14 hours of fasting by a laboratory technician. Following the collection of the blood samples, the plasma will be separated from the blood cells, which will then be separated from one another using a Ficoll solution. The plasma and PBMC samples will be stored in microtubes in a freezer at -80°C until the requisite tests have been conducted. The concentrations of plasma lipids will be determined using standard kits. LBP concentrations will be quantified using enzyme-linked immunosorbent assay (ELISA) kits. Total RNA will be extracted from the PBMC samples and cDNA will be synthesized using a cDNA synthesis kit. Subsequently, the expression of the GPR109A and GPR43 genes will be quantified through the use of specific primers and a quantitative PCR assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of coronary heart disease who have recently undergone coronary angioplasty

Exclusion Criteria:

* End-stage renal disease
* Inflammatory bowel syndrome (IBD),
* Recent glucocorticoid or antibiotic treatment,
* Cancer undergoing chemotherapy or radiotherapy,
* Any alteration to the treatment plan, including changes in drug type or surgical intervention

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Plasma lipids | At the beginning of the study and two months later
  Plasma concentrations of triglyceride, cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol
Plasma inflammatory biomarkers | At the beginning of the study and two months later
  Plasma c-reactive protein, Interleukin-6, ICAM-1, and VCAM-1
Plasma lipopolysaccharide-binding protein | At the beginning of the study and two months later
  Plasma concentrations of lipopolysaccharide-binding protein

SECONDARY OUTCOMES:
Fecal bacteria | At the beginning of the study and two months later
  Relative abundance of certain bacteria in feces
Expression of GPR43 and GPR109A | At the beginning of the study and two months later
  The expression of the GPR109A and GPR43 genes in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Shahid Modaress Hospital, Tehran, Tehran Province
  - Shahid Modarres Hospital, Tehran, Tehran Province

IPD SHARING:
Plan to Share IPD: Undecided